CLINICAL TRIAL: NCT00912665
Title: Regulation of Optic Nerve Head Blood Flow During Combined Changes in Intraocular Pressure and Arterial Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Ass.Prof.Priv.Doz.Dr., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OPHT-150808
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Healthy
Keywords: Optic Nerve Head Blood Flow; Intraocular Pressure; Regional Blood Flow; Ocular Physiology; Optic Disk
MeSH Terms: interventions — Laser-Doppler Flowmetry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Healthy Volunteer (Experimental)
  Interventions: Device: Laser Doppler Flowmetry; Device: Goldmann applanation tonometer; Other: squatting; Device: Suction cup

INTERVENTIONS:
Device: Laser Doppler Flowmetry — blood flow measurements at the temporal neuroretinal rim to assess optic nerve head blood flow
Device: Goldmann applanation tonometer — intraocular pressure measurements
Other: squatting — Subjects will perform squatting for 6 minutes while either blood flow or intraocular pressure measurements
Device: Suction cup — Experimental stepwise increase of intraocular pressure while either optic nerve head blood flow or intraocular pressure measurements

SUMMARY:
Autoregulation is defined as the ability of a vascular bed to adapt its vascular resistance to changes in perfusion pressure. In the eye, several studies have reported that retinal blood flow is autoregulated over a wide range of ocular perfusion pressures. In the optic nerve head only few data are available. Large scale studies have shown that reduced ocular perfusion pressure is an important risk factor for the prevalence, the incidence and the progression of primary open angle glaucoma.

Former studies that investigated ocular blood flow autoregulation only measured choroidal blood flow. For the optic nerve head only few data are available, although it seems likely that it underlies similar autoregulatory mechanisms.

The primary goal of the present study is to gain more insight into these phenomena in humans.

The present study aims to investigate the pressure/flow relationship as a measure for optic nerve head autoregulation during combined changes of intraocular pressure and arterial pressure. Intraocular pressure will be increased by the use of a suction cup technique, mean arterial pressure will be increased by squatting. During the whole procedure, optic nerve head blood flow will be measured continuously.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 35 years, nonsmokers
* Men and women will be included in equal parts
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal findings in the laboratory testings unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia less than 1 diopter

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug (except oral contraceptives)
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Blood donation during the previous 3 weeks

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Optic nerve head pressure-flow relationship | in total 3x on 2 study days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Vienna, Austria